CLINICAL TRIAL: NCT05791656
Title: Composite Interference Screw in the Surgical Reconstruction of Knee Cruciate Ligaments: a Prospective Observational Study
Brief Title: Interference Screw Mectascrew-C Postmarket Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P07.001.09
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Injuries; Posterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Mectascrew-C — reconstruction of ACL or PCL rupture

SUMMARY:
An observational prospective study with the aim to analyze the presence at 6 months of a specific composite IS (Medacta Mectascrew C) in the reconstructive treatment of ruptured ACL or PCL by means of an autograft or allograft.

DETAILED DESCRIPTION:
This is an observational prospective study with the aim to determine the presence of the composite IS (Mectascrew-C) at 6 months following ACL or PCL reconstruction.

Patients with an ACL or PCL tear scheduled for surgery at one of the EOC's hospitals will be enrolled in the study, after the subscription of informed consent. The injured ligament will be restored with an auto- or allograft that will be fixed with a composite IS (Mectascrew-C, 70% PLDLLA, 30% β-TCP, Medacta International SA).

The data will be collected from patient's medical histories (data about diagnosis, patients' characteristics and surgery) and after operation, during the orthopaedic follow-up visits, planned at 1, 3 and 6 months, in order to assess the functional outcomes (IKDC objective and subjective) and the knee stability (ROM, Pivot Shift or Reverse Pivot Shift test, anterior or posterior drawer test) of the patients.

The treated knee will be also evaluated radiologically with an MRI at 6 months to assess the IS reabsorption. The results of this exam will be correlated to the pre-operative findings and to the functional and clinical outcomes evaluated with the different forms

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 16-60 yrs
* Pre-operative MRI confirming the ACL or PCL rupture
* Scheduled for surgical reconstruction of ACL or PCL
* BMI>18 and <35 kg/m2
* Ability to give informed consent by signature

Exclusion Criteria:

* Age under 16 or over 60 yrs
* Degenerative osteopathies
* Local bone tumors
* Deformities of the bone, or general conditions of the bone, which preclude the implantation in the opinion of a physician
* Systemic diseases and metabolic disorders that may compromise the outcome of the surgery

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with an ACL or PCL rupture, and meeting the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Interference screw presence | 6 months
  via MRI imaging at 6 months after surgery, the presence of the Mectascrew-C will be assessed

SECONDARY OUTCOMES:
Mobility outcomes evaluation | 1, 3 and 6 months
  Assessment throught Range Of Motion of operated knee calculated as degree
Functional outcomes evaluation | 1, 3 and 6 months
  Assessment throught IKCD score. a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Knee stability evaluation of ACL intervention | 1, 3 and 6 months
  Pivot shift test. A positive test indicate an injury at ACL
ACL integrity assessment | 1, 3 and 6 months
  Anterior drawer test. An anterior translation more than 6 mm indicate a positive test with injuried ACL
Knee stability evaluation of PCL intervention | 1, 3 and 6 months
  Reverse Pivot Shift test. In the presence of a posterolateral injury with the knee flexed, the tibia follows gravity and drops into posterolateral subluxation (positive Reverse Pivot Shift Test).
PCL integrity assessment | 1, 3 and 6 months
  Posterior drawer test. The test is considered positive if there is a lack of end feel or excessive posterior translation.
Device safety evaluation | 1, 3 and 6 months
  collection of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, Prof Med, Principal Investigator — EOC , Service of Orthopaedics and Traumatology, Lugano (Switzerland)
Locations (1):
- EOC, Service of Orthopaedics and Traumatology, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No